CLINICAL TRIAL: NCT05304299
Title: Alleviating Effects Against High Intraocular Pressure by Oral Intake of Cordyceps Cicadae Mycelia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Han-Hsin Chang (Other)
Collaborators: Grape King Bio Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Han-Hsin Chang, Principal Investigator, Chung Shan Medical University
Organization: Chung Shan Medical University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB-19-024
Record Dates: First submitted 2022-03-04; First posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Supplement

STUDY DESIGN:
Intervention Model Description: Two groups of subjects are subject to pre-test and post-test intraocular pressure measurements.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cordyceps Cicadae Mycelia only (Experimental): Only Cordyceps Cicadae Mycelia will be given.
  Interventions: Dietary Supplement: Cordyceps Cicadae Mycelia
- Cordyceps Cicadae Mycelia with Taflotan (saflutan) (Experimental): Cordyceps Cicadae Mycelia with Taflotan (saflutan) will be given.
  Interventions: Dietary Supplement: Cordyceps Cicadae Mycelia

INTERVENTIONS:
Dietary Supplement: Cordyceps Cicadae Mycelia — Cordyceps Cicadae Mycelia will be given to test its potential for alleviation of high intraocular pressure.

SUMMARY:
This study will investigate the effects of lowering intraocular pressure by oral intake of Cordyceps cicadae mycelia, to provide evidence-based data for high intraocular pressure relief.

DETAILED DESCRIPTION:
Study purpose This study investigated the effeicacy of oral Cordyceps cicadae mycelia for the relief of high intraocular pressure.

Subjects

1. The total recruitment of subjects is 60 people, aged between 20 to 75 years.
2. Subjects with intraocular pressure more than or equal to 21 mmHg are included, irrespective of whether on us of Taflotan (saflutan).

Methods

1. Informed consents will be obtained from subjects first. The subjects with pre-test intraocular pressure over or equal 21 mm Hg are advised to orally take two capsules containing a total of 500 mg of Cordyceps cicadae mycelia. After 90 minutes, the subjects are evaluated for intraocular pressure.

The pre-test and and post-intake intraocualr pressure and blood pressure data will be compared by paired t test for significant differences if any.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 20 and 75 years old, regardless of gender.
2. Pre-test confirmation of high intraocular pressure.
3. Subjects should understand the trial and agree to join the project.

Exclusion Criteria:

1. Age under 20 or over 75 years.
2. Use intraocular pressure lowering drugs other than Taflotan (saflutan).
3. Using beta-blockers or diuretics.
4. Being pregnant.
5. Disabled individuals with specific diseases or malfunction, for example tumours at terminal stage, blindness.
6. Loss of self-consciousness and behavioral capacity.
7. Patients with major diseases.

Withdrawal criteria All subjects may withdraw at any time without any reason. The act of withdraw does not affect rights for them to seek medical advice or treatments.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure | 0 minutes (before given Cordyceps Cicadae Mycelia)
  Intraocular pressure of both eyes will be assessed
Intraocular pressure | 90 minutes after given Cordyceps Cicadae Mycelia
  Intraocular pressure of both eyes will be assessed
Blood pressure | 0 minutes (before given Cordyceps Cicadae Mycelia)
  Both systolic and diastolic blood pressures will be assessed
Blood pressure | 90 minutes after given Cordyceps Cicadae Mycelia
  Both systolic and diastolic blood pressures will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Han-Hsin Chang, PhD, Principal Investigator — Chung Shan Medical University
Locations (1):
- Han-Hsin Chang, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No